CLINICAL TRIAL: NCT02793531
Title: Assessment of Anabolic Responsiveness to Protein Intake in Advanced Cancer
Brief Title: Anabolic Response Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment potential in local community
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2015-0460
Record Dates: First submitted 2016-05-24; First posted 2016-06-08 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy matched controls (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed. Subjects may sign a medical release form to obtain medical and psychological information about them that will help determine study eligibility or can be used for later coding.
  study day: muscle mass and function tests, resting energy expenditure, stable isotope infusions with blood draws, and questionnaires regarding quality of life, mood and depression, diet.
  Interventions: Other: Stable isotope amino acid infusion
- Cancer subjects (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed. Subjects may sign a medical release form to obtain medical and psychological information about them that will help determine study eligibility or can be used for later coding.
  study day: muscle mass and function tests, resting energy expenditure, stable isotope infusions with blood draws, and questionnaires regarding quality of life, mood and depression, diet.
  Interventions: Other: Stable isotope amino acid infusion

INTERVENTIONS:
Other: Stable isotope amino acid infusion — such as glycerol, D2O, tyrosine, phenylalanine, glucose, arginine, and citrulline

SUMMARY:
Weight loss and muscle wasting commonly occurs in patients with cancer, negatively influencing their quality of life, treatment response and survival. Weight changes in patients with cancer may be the consequence of energy imbalance and disturbances in protein metabolism, poor treatment tolerance, hormonal alterations, systemic inflammation etc. This results in body composition modifications in favor of fat gain and/or lean body mass loss in early stage cancer. However, in advanced cancer mostly loss of both fat mass and lean mass has been found.

Unfortunately, gains in muscle mass are difficult to achieve. In a previous study of the Investigators, a bolus (15 g) of an essential amino acid mixture as present in milk protein was able to stimulate whole-body protein anabolism equally and effectively in weight-losing patients with lung cancer. This indicates the high potential of proteins with high essential amino acids as therapeutic agents to increase muscle mass in these patients. However, the dose-response effect to reach optimal whole-body protein anabolism is yet unknown and can differ among patients. Therefore, the Investigators would like to study the effects of several dosages of a protein with high essential amino acid levels, administered by sip feeding, on whole-body protein anabolism in patients with cancer in comparison with healthy older adults. Furthermore, the individual protein requirements of cancer patients may be established as this is the cornerstone of nutritional support. Specifically to establish 'the anabolic threshold', when protein breakdown equals synthesis and the response and the relation between protein intake and net protein synthesis are critical.

DETAILED DESCRIPTION:
In this study, the Investigators will test the following hypothesis: A protein meal with high EAA levels will stimulate protein anabolism in a dose-dependent way but the exact relationship differs among cancer patients. The primary endpoint will be the extent of stimulation of net whole-body protein synthesis at each level of protein intake in the individual cancer and control subject. This project will provide important clinical information on the anabolic capacity of dietary protein with high EAA levels and the level of protein intake required to become anabolic in cancer patients on an individual bases. In this way, this study will provide preliminary data for the development of individualized nutritional strategies that will stop the process of ongoing muscle loss in cancer patients.

General aims:

* To study the whole-body protein anabolic effect of several dosages of a high-quality protein sip feeding in cancer subjects as compared to healthy controls.
* To investigate the anabolic threshold in subjects with cancer as compared to healthy controls.

The mechanisms underlying lean tissue loss in cancer remain to be unraveled, which may be because of the complexity of the metabolic alterations that are present when symptoms such as weight loss become obvious. Multiple factors like anorexia and inflammation are present in cancer, all contributing to the loss of lean tissue in these patients by creating a drain on the body protein stores. Previous studies showed that oral supplementation of large amounts of calories in cancer is only partially successful and this indicates that the composition of dietary supplements and meals is important to successfully counteract muscle wasting. Although our previous study supports the concept of supplementing high-quality milk proteins in lung cancer subjects, the dose-response anabolic effects of proteins with high EAA levels are still unclear. Furthermore, there is no insight in the actual protein requirements in cancer. The knowledge gained from this study will benefit our insight in terms of promotion of protein gain after feeding in cancer patients.

ELIGIBILITY:
Inclusion criteria cancer subjects:

* Age 18 years or older
* Ability to lie in supine or elevated position for 8 hours
* Diagnosed with stage III/IV cancer (all solid tumors excluding breast or prostate)
* No chemotherapy/radiotherapy within past month prior to the study day
* Willingness and ability to comply with the protocol

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Age 18 years or older
* Ability to lay in supine or elevated position for 8 hours
* No diagnosis of cancer
* No diagnosis of diabetes
* Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only)
* Presence of fever within the last 3 days
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* BMI of < 18.5 or ≥ 35 kg/m2 (for healthy control group only)
* Dietary or lifestyle characteristics: Current alcohol or drug abuse, Use of protein or amino acid containing nutritional supplements within 5 days prior to the study day
* Known allergy to milk or milk products
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in net whole-body protein synthesis | 0, 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 225, 240, 260, 280, 300, 320, 340, 360 ± 5 min
  Change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Body Composition | 15 minutes on screening or study day 1
  Body composition as measured by Dual-Energy X-ray Absorptiometry
Skeletal muscle strength | on study day 1
  handgrip
Skeletal muscle strength | on study day 1
  kin-com 1-leg test
Respiratory muscle strength | on study day 1
  Maximum inhalation and exhalation pressure
Gut function | In postabsorptive and prandial state every 20 minutes up to 6 hours before each sip feeding on study day
  Digestion of the stable tracers of amino acid
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS) | Postabsorptive state during 3 hours and change after feeding on study day 1
  a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Group differences in activity as measured by Physical Activity Scale for the Elderly (PASE) | Postabsorptive state during 3 hours and change after feeding on study day 1
  questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
Group differences in state of mood as measured by the Profile of Mood State (POMS) | Postabsorptive state during 3 hours and change after feeding on study day 1
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment. Healthy populations take 3 to 7 minutes to complete, and others may take up a bit longer.
appetite questionnaire | study day 1
  The subject is asked to rate various aspects of their appetite as relates to overall health
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT) | Postabsorptive state during 3 hours and change after feeding on study day 1]
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT) | Postabsorptive state during 3 hours and change after feeding on study day 1
  The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonetic verbal fluency. The raw score (total and mean words recorded across the three trials) was reported.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | Postabsorptive state during 3 hours and change after feeding on study day 1
  assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in attention and executive functions as measured by Brief-A | Postabsorptive state during 3 hours and change after feeding on study day 1
  a standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
diet recall | Postabsorptive state during 3 hours and change after feeding on study day 1
  The subject is asked to recall in detail all the food and drink consumed during the 24 hours prior to the test day.
Group differences in attention and executive functions as measured by Trail Making Test (TMT) | Postabsorptive state during 3 hours and change after feeding on study day 1
  Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Functional Status | Postabsorptive state during 3 hours and change after feeding on study day 1
  Functional status will be assessed by the Karnofsky Performance Score, a widely used method to assess the functional status of a cancer patient. It describes a patient's functional status as a comprehensive 11-point scale ranging from 0% to 100%.
Group differences in learning and memory as measured by Auditory Verbal Learning Test (AVLT) | Postabsorptive state during 3 hours and change after feeding on study day 1
  a verbal episodic memory test that evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, retention and recognition of information.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No